CLINICAL TRIAL: NCT06894576
Title: Development of a Risk Stratification Score for Recurrent Venous Thromboembolism and Treatment-related Clinically Relevant Bleeding in Patients With Cancer-associated Thrombosis
Acronym: CAN-CATCH
Status: Recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20240308-01T
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cancer-associated Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma from citrated whole blood, whole blood, plasma from whole EDTA blood tubes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to prospectively develop a risk assessment model (RAM) that accurately identifies anticoagulated cancer-associated thrombosis (CAT) patients at low- and high-risk of recurrent venous thromboembolism (VTE) and clinically relevant bleeding within 6 months following the CAT diagnosis and to create a biobank of plasma and whole blood samples for further translational research in cancer genetics and hemostasis.

DETAILED DESCRIPTION:
CAN-CATCH study is a prospective cohort study to develop a risk assessment model for VTE recurrence and clinically relevant bleeding in patients with CAT. The study is anticipated to recruit for a period of 2 years with a 3-year completion timeline.

The primary objective of this study is to prospectively develop a RAM that accurately identifies anticoagulated CAT patients at low- and high-risk of CAT recurrence and clinically relevant bleeding within 6 months following the CAT diagnosis.

The secondary objective is to create a biobank of plasma and DNA samples at the time of CAT diagnosis, linked to the annotated dataset for future translational biomarker research in cancer genetics and hemostasis.

At approved sites, participants will donate 4x4.5 mL 3.2% citrate tubes and 3x10 mL ethylenediaminetetraacetic (EDTA) tubes for blood banking.

In addition to the initial enrollment visit, participants that are enrolled will have a follow up at day 90 ± 14 days (3 months) and at day 180 ± 14 days (6 months) from randomization. Post enrollment follow-up visits will include assessment and documentation of any major and clinically relevant non-major bleeding (CRNMB), investigations for VTE, change in cancer treatment regimen, VTE risk factors, bleeding risk factors and death. Participants who experience an outcome event should continue to be followed

ELIGIBILITY:
Inclusion Criteria:

* Objectively documented distal and/or proximal DVT of the limb (upper or lower extremity) and/or PE, splanchnic vein thrombosis and/or cerebral sinus vein thrombosis in presence of active cancer of all types
* Intended treatment of CAT for at least 6 months with parenteral or oral anticoagulants at therapeutic dosing.
* Estimated life expectancy > 6 months
* Willingness to give an informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Unusual site CAT (gonadal vein thrombosis, ovarian vein thrombosis, retinal vein thrombosis)
* Superficial vein thrombosis
* Refusal of informed consent > 72 hrs of anticoagulants
* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cancer Associated Thrombosis receiving anticoagulation treatment with a follow-up of 6 months
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recurrent VTE | 6 months
  The primary outcome of the study will include objectively confirmed recurrent VTE (distal and/or proximal deep vein thrombosis (DVT) and/or pulmonary embolism (PE) and/or splanchnic vein thrombosis and/or cerebral venous sinus thrombosis

SECONDARY OUTCOMES:
Overall mortality | 6 months
  Post-enrollment follow-up visits will include documentation of death if occuring at any time during the 6 month follow up period
Clinically relevant bleeding | 6 months
  Post-enrollment follow-up visits will include assessment and documentation of any major and CRNMB and bleeding risk factors at any time during the 6 month follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Carrier, MD, Principal Investigator — Ottawa Hospital
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada